CLINICAL TRIAL: NCT03589898
Title: Imaging Biomarkers of Social Cognition and Pharmacologic Target Engagement in Autism Spectrum Disorder
Brief Title: Study of Neuroimaging Biomarkers of Social Cognition Deficits in Adolescents (Age 13-17) With Autism Spectrum Disorder and Effects of Gabapentin
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, David Cochran, Assistant Professor of Psychiatry and Pediatrics, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H00012656; 1K23MH113008-01A1 (NIH)
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Autism Spectrum Disorder
Keywords: magnetic resonance imaging; spectroscopy; GABA; glutamate; social cognition
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gabapentin (Experimental): Single dose of gabapentin 900 mg will be given and neuroimaging markers will be measured before and after administration of gabapentin
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Single dose of gabapentin 900 mg

SUMMARY:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder that is increasing in prevalence, and is characterized by deficits in social communication and interaction across multiple contexts, and restricted, repetitive patterns of behavior, interests, or activities. The majority of individuals with ASD have poor outcomes in the area of social functioning; however, there are no medical treatments available that target the core social communication deficits. The goal of the proposed research is to understand the neurobiological role of an imbalance in excitatory (glutamate) and inhibitory (gamma-aminobutyric acid, GABA) neurotransmission in the social cognition deficits in ASD, and to develop proton magnetic resonance spectroscopy as a measurement of target engagement to measure the ability of a medication, gabapentin, to increase cortical GABA levels. Spectrally-edited proton magnetic resonance spectroscopy (1H-MRS) provides an ideal method for measuring cortical GABA levels. All proposed studies will be in 70 adolescents (male and female) with ASD (age 13 to 17 years). Specific Aim 1: To measure correlations of 1H-MRS GABA levels in the anterior cingulate cortex (ACC) and occipital cortex (OC) with clinical measures of social cognition at baseline. Specific Aim 2: To measure the effect of an initial one time dose of gabapentin on 1H-MRS GABA levels in the ACC and OC. The hypotheses are 1) that higher social cognition ability will be positively correlated with GABA in the ACC but not in the OC (a control, non-social cognition-related region) of individuals with ASD, and 2) that gabapentin will increase GABA levels in the ACC and OC of youth with ASD.

DETAILED DESCRIPTION:
The investigators will complete a 1H-MRS study in 42 adolescents with ASD. Given the low burden on patients, it is assumed that 90% of those recruited to participate in baseline 1H-MRS (Aim 1) will also consent/assent to repeated 1H-MRS after gabapentin administration (Aim 2). Projections from the preliminary study were used to select a proposed number of subjects that would be both achievable in the time frame of study and adequate to evaluate the research hypotheses.

Psychiatric comorbidity will be assessed based on DSM-5 criteria by clinical interview and administration of the Kiddie-Schedule for Affective Disorders and Schizophrenia (Present and Lifetime version; K-SADS-PL).

T1- and T2-weighted high resolution structural imaging (T1- and T2-weighted (MPRAGE)) will be acquired. These structural MRI scans will be analyzed using FreeSurfer (Martinos Center for Biomedical Imaging, Charlestown, MA) and Statistical Parameter Mapping (SPM8-http://www.fil.ion.ucl.ac.uk/spm/software/spm8/) to determine white matter, gray matter and CSF contributions to the MRS voxel for partial volume correction. This data will be analyzed for variation with age, and used as a co-variate in the statistical analysis plan.

MRS data will be acquired from the Anterior Cingulate Cortex and Right anterior insula. Imaging sessions will be conducted at the Advanced MRI Center (AMRIC) at UMMS, which houses a 3.0 Tesla Philips Achieva MRI research scanner (Philips Healthcare, Best, Netherlands) and 32-channel phase-array receiver SENSE head coil. AMRIC is dedicated to research and the MRI system has considerable evening and weekend availability. A Board certified neuroradiologist associated with the AMRIC at UMMS reviews all MRI scans. In the event of an unexpected, clinically important finding, the primary investigator will be informed. The investigator will share the finding with the participant and be in contact with the participant's primary care physician (PCP) in order to help decide the appropriate follow-up care/work up that is needed (consent will be obtained to contact each child's PCP during the study consent process).

GLU+GLN absolute levels will be quantified, and GABA levels will be quantified using the total creatine (tCr) peak as a reference. Macromolecule-suppressed editing will be used with MEGA-PRESS sequence, including prospective frequency correction to address the impact of drift and motion during scans.

Neurotransmitter levels will be correlated with social cognition measures. In females of reproductive age, menstrual cycle charting will be done for 2 months prior to scan, and imaging will be timed to target the mid-luteal phase, as cortical GABA levels fluctuate during the menstrual cycle and are most similar to levels in males during the luteal phase. In analysis of female subject data, menstrual phase will be confirmed on the day of the scan by measurement of serum estradiol and progesterone levels, and these levels will be used as covariates in the analysis. Exploratory analysis will be used to seek correlations with all clinical measures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 13-17 years
2. English as primary language (both child and legal guardian)
3. DSM-5 criteria for Autism Spectrum Disorder
4. IQ >70 per Weschler Abbreviated Scale of Intelligence (WASI)
5. Informed assent for the study (The guardian must also give written informed consent).

Exclusion Criteria:

1. Any neurological disorder (e.g., cerebral palsy, fetal alcohol syndrome, cerebral neoplasm, bacterial meningitis, epilepsy, etc.)
2. Genetic disorders (e.g., Fragile X, Rett Syndrome, etc.)
3. Preterm (<36 weeks)
4. Failure to thrive within first year of life
5. Contraindications for MRI, such as metallic or electronic implants in the body, or severe claustrophobia
6. History of head trauma with loss of consciousness for more than 30 minutes
7. Unstable psychiatric illness, history of psychotic disorder, or psychiatric illness that would prevent the subject from being able to complete study protocol
8. Unstable medical illness such as diabetes, asthma, thyroid disease.
9. Currently on medications that cause respiratory depression, e.g. opioids, benzodiazepines
10. Clinically significant suicidal ideation at screening as assessed by the Columbia Suicide Severity Rating Scale
11. IQ < 70
12. History of intolerance to gabapentin or pregabalin
13. Current substance use (including nicotine)
14. Pregnancy at time of 1H-MRS or gabapentin administration
15. Current treatment with gabapentin
16. History of Renal Dysfunction
17. Subjects who weigh less than 36 kg
18. Subjects who weigh more than 105.8 kg

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Cortical GABA in Anterior Cingulate Cortex | 6 hours post-administration
  Cortical gamma-aminobutyric acid levels measured using magnetic resonance spectroscopy with voxel placed in bilateral anterior cingulate cortex
Cortical GABA in Right Anterior Insula | 6 hours post-administration
  Cortical gamma-aminobutyric acid levels measured using magnetic resonance spectroscopy with voxel placed in right anterior insula

SECONDARY OUTCOMES:
Cortical Glx in Anterior Cingulate Cortex | 6 hours post-administration
  Cortical glutamate/glutamine levels measured using magnetic resonance spectroscopy with voxel placed in bilateral anterior cingulate cortex
Cortical Glx in Right Anterior Insula | 6 hours post-administration
  Cortical glutamate/glutamine levels measured using magnetic resonance spectroscopy with voxel placed in right anterior insula

CONTACTS AND LOCATIONS:
Overall Officials: David Cochran, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Plan for sharing individual participant data is still being discussed and developed by study team.